CLINICAL TRIAL: NCT03842293
Title: Clinical Evaluation of PROMIS Pediatric Person Reported Outcome Measures in Children With Chronic Kidney Disease
Brief Title: Clinical Evaluation of PROMIS in CKD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-013723; 1U19AR069525 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the clinical validity of a set of PROMIS pediatric person-reported outcome measures in patients with chronic kidney disease. The evaluation includes longitudinal assessments of how measures change in association with clinical changes.

DETAILED DESCRIPTION:
The National Institutes of Health (NIH)-sponsored Patient-Reported Outcomes Measurement Information System (PROMIS) network has developed over 20 pediatric instruments, both child-report and parent-proxy editions. Cross-sectional evaluations of the validity of the instruments have established that they are ready for integration into clinical research and practice. The next step in their ongoing evaluation is to assess their prospective clinical validity in a variety of health conditions. This study addresses the clinical evaluation of the measures in children with chronic kidney disease (CKD).

Through baseline surveys and six follow-up surveys over a two-year period, Investigators are collecting self-report (child) and parent-proxy report of 11 pediatric PROMIS measures. Each of these PROMIS measures is described in the Main Outcome Measures section. Investigators are also collecting assessments of disease activity from clinical data. The selection of self-report and parent proxy patient-reported outcome (PRO) measures were determined through qualitative content validation. The analytic goal of this project is to evaluate baseline (cross-sectional) and longitudinal associations between PROMIS pediatric outcome measures and changes in the clinical status of patients with CKD. Our primary hypothesis is that as kidney function declines, self-reported health will worsen.

ELIGIBILITY:
Inclusion Criteria:

* Child is 8-21 years old at time of enrollment
* Child is a Chronic Kidney Disease in Children (CKiD) patient OR a child who receives pediatric nephrology care at a CKiD site that participates in PEDSnet, a national pediatric learning health system
* Child seen by a pediatric nephrologist in the past 24 months
* Child has two eGFR readings (computed from serum creatinine) between 6-89 ml/min at least 3 months apart (eGFR of this level indicates CKD)
* Child speaks English
* Parent is the parent or legal guardian for the child
* Parent speaks English

Exclusion Criteria:

* Child is currently receiving dialysis
* Child received a kidney transplant
* Child has a parent-reported cognitive limitation that would preclude them from completing a questionnaire
* Child does not speak English
* Parent does not speak English
* Parent is not the parent of legal guardian for the child

Ages: 8 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants were initially recruited through an existing study, the Chronic Kidney Disease in Children (CKiD) study. CKiD is a long-term prospective cohort study that currently follows 364 children with CKD from 54 North American centers. Recruitment was expanded to also enroll children between the ages of 8 and 21 years who had been seen at a nephrology clinic at two CKiD participating sites, Children's Hospital of Philadelphia (CHOP) and Cincinnati Children's Hospital and Medical Center (CCHMC) and had two eGFR readings (computed from serum creatinine) between 6-89 ml/min at least 3 months apart (eGFR of this level indicates CKD).
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in sleep disturbance | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 8 items from PROMIS sleep-related disturbance domain. Participants rate their experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in sleep-related impairment | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 4 items from PROMIS sleep-related impairment domain. Participants rate their experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in fatigue | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 8 items from PROMIS fatigue domain. Participants rate their experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in life satisfaction | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 4 items from from PROMIS life satisfaction domain. Participants rate their experience using a five point scale ranging from not at all to quite a bit. Answers are converted to a t-score to compare to the general population.
Longitudinal change in meaning and purpose | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 4 items from from PROMIS meaning and purpose domain. Participants rate their experience using a five point scale ranging from not at all to quite a bit. Answers are converted to a t-score to compare to the general population.
Longitudinal change in psychological stress experiences | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Child self-report of 4 items from from PROMIS psychological stress experiences domain. Participants rate their experience using a five point scale ranging from not at all to quite a bit. Answers are converted to a t-score to compare to the general population.
Longitudinal change in global health | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Parent proxy report of 7 items from from PROMIS global health domain. Parents rate their child's experience using a five point scale ranging from poor to excellent. Answers are converted to a t-score to compare to the general population.
Longitudinal change in depressive symptoms | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Parent proxy report of 4 items from from PROMIS emotional distress - depressive symptoms domain. Parents rate their child's experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in anxiety | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Parent proxy report of 4 items from from PROMIS emotional distress - anxiety domain. Parents rate their child's experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in positive affect | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Parent proxy report of 4 items from from PROMIS positive affect domain. Parents rate their child's experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.
Longitudinal change in family relationships | Baseline and 3 month, 6 month, 12 month, 15 month, 18 month and 24 month follow-ups.
  Parent proxy report of 4 items from from PROMIS family relationships domain. Parents rate their child's experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Furth, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (16):
- United States (15):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - University of Michigan, Mott Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Levine Children's, Charlotte, North Carolina
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hopsital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada